CLINICAL TRIAL: NCT05003128
Title: Changes in Tear Lipid Layer Thickness After Short Exposure to Light Emitting Diode Displays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A-ER-108-489
Record Dates: First submitted 2021-07-29; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Lipid Tear Deficiency (Disorder); Dry Eye Disease
Keywords: Computer vision syndrome; Dry eye disease; Light emitting diode; Lipid layer thickness; Video display terminals
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LED screen (Experimental)
  Interventions: Device: LED screen (InnoLux, Taiwan)

INTERVENTIONS:
Device: LED screen (InnoLux, Taiwan) — Participants watch a short movie on an LED screen (InnoLux, Taiwan) for 15 minutes in a bright room. The viewing distance was approximately 1.5 meters.

SUMMARY:
Video display terminals (VDTs) are ubiquitous, and engagement in digital screens has grown substantially across all age groups worldwide. Prolonged exposure to VDTs is associated with the development of various health problems. By now, it is unclear whether transient exposure to VDTs leads to ocular surface changes, especially regarding lipid layer thickness (LLT). This study aim to determine if short-term exposure to light-emitting diodes (LEDs) leads to ocular parameter changes.

This is a prospective, cross-sectional study. Patients were recruited at the National Cheng-Kung University Hospital, a tertiary referral center in southern Taiwan, for examination, including best-corrected visual acuity (BCVA), intraocular pressure (IOP), lipid layer thickness (LLT), and blink rates and patterns before and after watching an LED display for 15 minutes. The estimated result is that the LLT and blink rates will decrease after VDT watching.

DETAILED DESCRIPTION:
Video display terminals (VDTs) are ubiquitous, and engagement in digital screens has grown substantially across all age groups worldwide. During the coronavirus disease 2019 (COVID-19) pandemic, lockdowns and increasing demand for digital learning and working have led to more frequent and sustained VDT use. Prolonged exposure to VDTs is associated with the development of various health problems, including psychosocial issues, venous thromboembolism, fatigue, and visual complaints.

Computer vision syndrome (CVS) is one of the most frequently encountered problems among VDT users. CVS comprises several visual and musculoskeletal symptoms resulting from VDT use, such as eye strain, dryness and burning sensation of the eye, blurred vision, and neck and shoulder pain. A major alteration is the development of dry eye disease (DED), occurring in 60 % of those with CVS. Dry eye symptoms, corneal erosions, short tear-film breakup time (BUT), low tear meniscus height, and meibomian gland dysfunction (MGD) are all DED presentations encountered by VDT users. The continuous use of VDTs is an established risk factor for CVS and DED. However, it is unclear whether transient exposure to VDTs leads to ocular surface changes, especially regarding lipid layer thickness (LLT).

This study investigated if the short-term use of light-emitting diode (LED) displays (one type of VDT) changed the ocular parameters, including best-corrected visual acuity (BCVA), intraocular ocular pressure (IOP), the CVS-Questionnaire (CVS-Q) score, the blink rate, the partial blink ratio, and LLT. To our knowledge, this is the first study to focus on the immediate effects of LEDs on the eye.

This prospective clinical study was conducted in the Ophthalmology Department of the National Cheng Kung University Hospital (NCKUH), Tainan, Taiwan. The study was approved by the Institutional Review Board of NCKUH and followed the tenets of the Declaration of Helsinki. Written informed consent was obtained from all the participants.

The inclusion criteria were generally healthy individuals aged between 20 and 65 years who were willing to participate in the study. The exclusion criteria were ages below 20 or over 65 years, a BCVA score of <0.1 on the Landolt C chart in either eye, a BCVA difference of >0.2 between the eyes, and a history of ocular diseases or previous ocular surgery.

Participants were instructed to fill out a basic information form, including their name, sex, age, and contact information. They were also informed to avoid wearing contact lenses for two days before the test. The experiment was conducted on August 22, 2020. For the baseline test, the participants were asked to complete the CVS-Q to assess their CVS. Next was a series of ocular examinations, including BCVA, IOP, LLT, an optical coherence tomography (OCT) scan of the macula, and fundus autofluorescence (FAF) imaging. The LLT and blink rates were measured using the LipiView II Ocular Surface Interferometer following the standard protocol (TearScience, Morrisville, NC, USA). After the examination, the participants watched a short movie on an LED screen (InnoLux, Taiwan) for 15 minutes in a bright room. The viewing distance was approximately 1.5 meters. After the movie ended, the participants were instructed to complete the CVS-Q and undergo the BCVA, IOP, and LLT tests again. The baseline BCVA, IOP, OCT, and FAF images of each participant were reviewed by three NCKUH ophthalmologists to screen for clinically significant ocular pathology.

Statistical analyses were performed using R software version 4.1.0 (R Core Team, Vienna, Austria) and SAS Enterprise Guide (version 9.4; SAS Institute Inc., Cary, NC, USA). Paired t-tests were used to compare the BCVA, IOP, CVS-Q score, LLT, blink rate, and the partial blink ratio before and after watching the LED display. Statistical significance was set at P <0.05.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy individuals aged between 20 and 65 years who were willing to participate in the study

Exclusion Criteria:

* ages below 20 or over 65 years
* a BCVA score of <0.1 on the Landolt C chart in either eye
* a BCVA difference of >0.2 between the eyes
* a history of ocular diseases or previous ocular surgery

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-22 (Actual); Study Completion 2020-08-22 (Actual)

PRIMARY OUTCOMES:
Lipid Layer Thickness | Change from baseline lipid layer thickness at 15 minutes

SECONDARY OUTCOMES:
Visual Acuity | Change from baseline visual acuity at 15 minutes
Intraocular Pressure | Change from baseline intraocular pressure at 15 minutes
Blink rates | Change from baseline blink rates at 15 minutes
Computer Vision Syndrome Questionnaire Score | Change from Baseline Computer Vision Syndrome Questionnaire Score at 15 minutes
  The Computer Vision Syndrome Questionnaire is a validated questionnaire to assess the severity of the computer vision syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hsun Huang, PhD, Study Chair — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The informed consent of this study specified that the participants' data would only be used in this study